CLINICAL TRIAL: NCT00353743
Title: A Randomized Clinical Trial on the Use or Not of Antibiotics After Hospital Discharge in Septic Abortion.
Brief Title: The Use of Antibiotics After Hospital Discharge in Septic Abortion
Acronym: APA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Rate of cure was higher than expected, IRB suspended for no additional benefit
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Ricardo Francalacci Savaris, HCPA-UFRGS
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 05-452; GPPG 05-452
Record Dates: First submitted 2006-07-13; First posted 2006-07-19 (Estimated); Last update posted 2008-12-19 (Estimated); Status verified 2007-03

CONDITIONS: Abortion, Septic
Keywords: infected abortion; treatment period; doxycycline; metronidazole; placebo
MeSH Terms: conditions — Abortion, Septic | interventions — Doxycycline; Metronidazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Patients that receive up to 10 days of doxycycline 200mg/day and metronidazole 500mg/day
  Interventions: Drug: doxycycline plus metronidazole
- 2 (Placebo Comparator): Patients that do not receive antibiotics, only placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: placebo — placebo
  Arms: 2
Drug: doxycycline plus metronidazole — doxycycline 200mg/day plus metronidazole 500mg/day up to 10 days of treatment (additional to the hospital treatment)
  Other Names: Vibramicina; Flagyl
  Arms: 1

SUMMARY:
The use of antibiotics in post-partum infection has been abbreviated. After 48 hours of clinical improvement, the patient is discharged from the hospital without antibiotics. No trials has been found in cases of septic abortion.

The purpose of the present study is to verify the need of antibiotics after clinical improvement in cases of septic abortion.

DETAILED DESCRIPTION:
Septic abortion is still a major cause of maternal mortality in developing countries. According to the WHO, 1 woman dies for every 270 illegal abortion (Ahman E, 2004). Infected abortion has an important role in maternal morbidity and mortality (Stubblefield PG, 1994). the diagnosis of infected abortion must be considered when a patient presents a history of delayed menses, vaginal bleeding, abdominal pain and fever (Brasil, 2000)

Prompt diagnosis and treatment are paramount steps to prevent complications. At Hospital de Clínicas de Porto Alegre, the use of gentamycin plus clindamicin before curettage is preconized (Savaris R, 2006). Nevertheless, the time of treatment it is not well established, varying from 7-14 days (Brasil, 2000).

A recent study with post-partum endometritis has shown that it is not necessary to extend the treatment to 14 days, after clinical improvement (Turnquest MA, 1998; French LM, 2004)

A randomized clinical trial comparing placebo with the standard protocol of treatment would define weather both treatments are equivalent or not.

Comparison: The prolonged use of antibiotics, after intravenous use of antibiotics and clinical improvement, will be compared to the use of placebo in cases of septic abortion.

Sample size and ethical issues The study protocol was approved by the ethics committee of Hospital de Clínicas de Porto Alegre.

To compare equivalence between the 2 treatments we calculated the sample size considering an alpha error of 0.05, a beta error of 0.1, and difference between the two groups of no more than 10%. We expected a 99% clinical cure with the standard protocol, and 95% for the alternative one. These figures yield a minimum of 42 patients in each group. Interim analysis will performed at 58 for possible early stopping, if clinical cure was < 95%, or for sample size re-estimation.

Randomization and treatment Subjects will be allocated in blocks of four at a time to create the allocation sequence. If the patient was eligible for the study, she will be allocated to one of the 2 treatments. The allocation will be concealed, coded and obtained from a central telephone number. Patients and those who assessed the outcomes were blind to group assignment. To avoid bias, both medications were manipulated by the hospital pharmacy and put in identically coded blisters and capsules.

Statistical analysis Student´s t-test, Mann-Whitney test, and Fisher´s exact test will be used for statistical analysis. The rates of cure were analyzed by "modified" intention to treat (Keech AC, 2003) and per protocol with 95% confidence intervals.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted at the hospital with a diagnosis of infected abortion and about to be discharged from the hospital.
* Use of intravenous antibiotics (gentamicin and clindamycin)
* Improvement of the clinical conditions for at least 48 hours (no fever, eating and walking normally, reduced vaginal bleeding)

Exclusion Criteria:

* Unwilling to participate in the study.
* Use of antibiotics previously within one week.
* Presence of tubo-ovarian abscess.
* Known allergy to doxycycline or metronidazole.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2006-05; Primary Completion 2007-11 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Clinical cure defined as no fever, no abdominal pain or bleeding. | 10 days after hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo F Savaris, MD, PhD, Principal Investigator — Hospital de Clínicas de Porto Alegre
Locations (1):
- Hospital de Clínias de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

REFERENCES:
- [Background] Ahman E, Shah I. Unsafe abortion: worldwide estimates for 2000. Reprod Health Matters. 2002 May;10(19):13-7. doi: 10.1016/s0968-8080(02)00012-5. PMID 12369316
- [Background] Stubblefield PG, Grimes DA. Septic abortion. N Engl J Med. 1994 Aug 4;331(5):310-4. doi: 10.1056/NEJM199408043310507. PMID 8022443
- [Background] Brasil.Ministério da Saúde. Abortamento infectado. In: Ministério da Saúde, ed. Urgências e emergências maternas: guia para diagnóstico e conduta em situações de risco de morte materna. 1 ed. Brasília: MS/FEBRASGO; 2000: 13-17.
- [Background] Savaris R. Abortamento. In: Freitas FM, Costa SMH, Lopes JG, eds. Rotinas em Obstetrícia. 5 ed. Porto Alegre: Artmed; 2006: 70-77.
- [Background] Turnquest MA, How HY, Cook CR, O'Rourke TP, Cureton AC, Spinnato JA, Brown HL. Chorioamnionitis: is continuation of antibiotic therapy necessary after cesarean section? Am J Obstet Gynecol. 1998 Nov;179(5):1261-6. doi: 10.1016/s0002-9378(98)70143-7. PMID 9822512
- [Background] French LM, Smaill FM. Antibiotic regimens for endometritis after delivery. Cochrane Database Syst Rev. 2004 Oct 18;(4):CD001067. doi: 10.1002/14651858.CD001067.pub2. PMID 15495005
- [Background] Heritier SR, Gebski VJ, Keech AC. Inclusion of patients in clinical trial analysis: the intention-to-treat principle. Med J Aust. 2003 Oct 20;179(8):438-40. doi: 10.5694/j.1326-5377.2003.tb05627.x. No abstract available. PMID 14558871
- See also: location of the study — http://www.hcpa.ufrgs.br